CLINICAL TRIAL: NCT03263013
Title: Non-invasive Intermittent Theta Burst Stimulation of the Dorsolateral Prefrontal Cortex in Patients With Functional Movement Disorders
Brief Title: Non-invasive Intermittent Theta Burst Stimulation of the Dorsolateral Prefrontal Cortex in People With Functional Movement Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170160; 17-N-0160
Record Dates: First submitted 2017-08-25; First posted 2017-08-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Movement Disorders
Keywords: Functional (BOLD) MRI
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FMD patients: patients with a diagnosis of clinically definite FMD who have been assessed at the HMCS clinic, and who have completed protocol 07-N-0190.

SUMMARY:
Background:

Functional movement disorder (FMD) causes involuntary movements, such as spasms, shaking, or jerks. These symptoms are not due to a recognized neurological or medical cause. Researchers want to better understand how the brain works to cause these symptoms.

Objective:

To test if intermittent theta burst stimulation (iTBS) affects brain areas involved in FMD symptoms. Also, to look at the effect of iTBS on mood and motor symptoms.

Eligibility:

Right-handed people ages 18-65 who have FMD and participated in protocol 07-N-0190

Design:

Participants will have 4 visits.

In Visit 1, participants will be screened with:

Medical history

Physical exam

Urine test

Questionnaires

Visit 1 might also include a brain MRI and functional MRI. The MRI scanner is a cylinder surrounded by a strong magnetic field. They will lie on a table that can slide in and out of the cylinder. For the functional MRI, they will be asked to perform tasks during the MRI scan.

Visit 2 will be 1-2 weeks after Visit 1. Visits 2, 3, and 4 will be no more than 48 hours apart. These include:

Electromyography: Small electrodes are taped to the skin. Muscle activity is recorded while participants receive magnetic stimulation of the brain.

Transcranial magnetic stimulation and iTBS: A wire coil is held on the scalp. A brief electrical current passes through the coil and creates a magnetic pulse to stimulate the brain. During iTBS, participants will sit quietly and watch a nature documentary. They will wear earplugs and a cap.

MRI

Functional MRI

Questionnaires

DETAILED DESCRIPTION:
Objectives:

The purpose of this protocol is to investigate feasibility and safety of intermittent theta burst stimulation (iTBS) targeting the left dorsolateral prefrontal cortex (DLPFC) in patients with functional movement disorders (FMD). We further aim at exploring whether iTBS of the DLPFC modulates amygdala activity, by investigating iTBS effects on resting-state fronto-amygdala connectivity and on amygdala BOLD response to valenced stimuli.

Study population:

FMD patients (N=6), aged 18-65 years, admitted at the Human Motor Control Section (HMCS) clinic, who have completed protocol 07-N-0190.

Design:

Participants will undergo four outpatient visits. On Visit #1 (baseline), patients will undergo a screening session to assess their eligibility to participate in the current study. They will undergo neurological and psychiatric assessment, as well as structural and functional magnetic resonance imaging. Intermittent TBS will be performed on three separated visits (Visit #2, #3 and #4; iTBS1, iTBS 2 and iTBS 3). During each visit, participants will receive three iTBS sessions over 1-hour, with a 15-minute interval between sessions. Each session will last 190 seconds and a total of 600 pulses will be delivered. Magnetic field intensity will be set at 120% of that participants observed daily resting motor threshold. The target will be identified using the neuronavigation system Brainsight. Following each iTBS visit, behavioral and functional imaging data will be collected.

Outcome measures:

Our primary outcomes will be to evaluate the safety and feasibility of different doses of iTBS of the left DLPFC in patients with FMD. In addition, in order to investigate amygdala engagement by DLPFC iTBS, the following exploratory outcomes will be analyzed: (1) Amygdala BOLD signal change in response to valenced stimuli, from baseline to iTBS3; (2) Amygdala BOLD signal change in response to valenced stimuli, from baseline to each timepoint (iTBS1- iTBS3), for each valence stimuli; (3) Change in fronto-amygdalar resting state functional connectivity, from baseline to iTBS3 (z-score); (4) Change in fronto-amygdalar resting state functional connectivity from baseline to each time point (iTBS1- iTBS3); (5) Change in the valence and arousal subjective levels, using the self-assessment Manikin, from baseline to each time point (iTBS1- iTBS3); (6) Correlations of percent amygdala BOLD signal change with changes in arousal and valence level; (7) Change in the scores on the simplified version of the FMD-RS from pre- to post treatment, for each timepoint.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of clinically definite functional movement disorder (as made by a neurologist)
* Ability to give informed consent
* Male and female participants between 18- 65 years of age
* Participation in protocol 07-N-0190
* Right handed (self-report)
* Ability to comply with all study procedures
* Abstinence from alcohol for at least 48 hrs prior to the study and caffeine on the day ofthe study (based on oral interview)

EXCLUSION CRITERIA:

* History of significant central nervous system disorders (primary or comorbid) such as neurodegenerative disorders, stroke, movement disorders, multiple sclerosis or epilepsy (clinical exam, MRI findings)
* History of psychotic disorder or bipolar disorder (clinical exam and/or SCID). Current acute mania and psychosis will also be excluded. As some degree of depressive symptoms is common in FMD patients, moderate unipolar depression will not be exclusionary (HAM-D score less than or equal to 18 will not be excluded)
* Current obsessive compulsive disorder (OCD) or post-traumatic stress disorder (PTSD)
* Active illicit substance use within the last 6 months (clinical exam and/or SCID).
* Current suicidal ideation (Columbia-Suicide Severity Rating Scale)
* Disease severity requiring inpatient treatment (clinical exam)
* Patients with movement symptoms at rest that may substantially inhibit resolution, comfort, or safety of MRI (clinical exam)
* Previous brain neurosurgery (self-reported history)
* History of head trauma that resulted in loss of consciousness for more than several seconds (self-reported history, TMS safety screening questionnaire, MRI findings)
* Regular use in the past 2 weeks of any of the following classes of medications: antiepileptics (except benzodiazepines, gabapentin and pregabalin), anti-parkinsonian medications, muscle relaxants, opiate medications and tricyclic antidepressants (selfreported history)
* Any history of seizures other than febrile childhood seizures (self-reported history)
* Family history of epilepsy (self-reported history, TMS safety screening)
* Patients with recurring fainting spells (self-reported history, TMS safety screening)
* Significant medical illness, including liver failure, kidney failure, congestive heart failure (clinical exam and/or medical records)
* Patients with documented hearing loss greater than or equal to 15dB at any frequency (medical records)
* Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the PI and after any consults if indicated, participation in the study is not in the best interest of the patient.
* Breastfeeding (self-report)
* NINDS employee/staff
* Subjects who have contraindications to MRI (we will follow the NMR Center guidelines for MR safety). Some of the exclusions are:

  * Have non-MRI compatible metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or ferromagnetic fragments in the eye or oral cavity as these make having an MRI unsafe.
  * Unable to lie flat on the back for the expected length of the experiment (50 minutes).
  * Have an abnormality on the brain imaging or neurologic examination not related to the diagnosis.
  * Uncomfortable being in a small space for the expected length of the experiment (50 minutes).
  * Non-removable body piercing or tattoo posing MRI risk
  * Pregnancy (urine pregnancy test)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FMD subjects will be recruited from patients assessed at the HMCS Clinic of NINDS/NIH, from the HMCS database, and from protocol 07-N-0190. Patients who have previously participated in protocol 07-N-0190 will be contacted over the telephone and offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
to evaluate the safety and feasibility of different doses of iTBS of the left DLPFC in patients with FMD. | throughout life of the protocol
  Percent of subjects experiencing adverse events (i.e., seizures, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stone J, Carson A, Duncan R, Roberts R, Coleman R, Warlow C, Murray G, Pelosi A, Cavanagh J, Matthews K, Goldbeck R, Sharpe M. Which neurological diseases are most likely to be associated with "symptoms unexplained by organic disease". J Neurol. 2012 Jan;259(1):33-8. doi: 10.1007/s00415-011-6111-0. Epub 2011 Jun 16. PMID 21674198
- [Background] Carson A, Stone J, Hibberd C, Murray G, Duncan R, Coleman R, Warlow C, Roberts R, Pelosi A, Cavanagh J, Matthews K, Goldbeck R, Hansen C, Sharpe M. Disability, distress and unemployment in neurology outpatients with symptoms 'unexplained by organic disease'. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):810-3. doi: 10.1136/jnnp.2010.220640. Epub 2011 Jan 21. PMID 21257981
- [Background] Gelauff J, Stone J, Edwards M, Carson A. The prognosis of functional (psychogenic) motor symptoms: a systematic review. J Neurol Neurosurg Psychiatry. 2014 Feb;85(2):220-6. doi: 10.1136/jnnp-2013-305321. Epub 2013 Sep 12. PMID 24029543
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0160.html